CLINICAL TRIAL: NCT02512796
Title: In Vitro Study of the Effect of Gadolinium Contrast on Fibrocytes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Other Study IDs: 18302
Record Dates: First submitted 2015-07-27; First posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Gadolinium Toxicity
Keywords: Liver transplantation; Renal transplantation; Pancreas transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Investigators plan to study the circulating fibrocytes numbers, changes in monocyte gene transcripts, identify polymorphism in gadolinium transport genes (OATPB1/3 and MRP2) and examine their osteogenic potential in cultures.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Transplant patients, MRI with Gadolinium contrast dye: Patients with kidney, pancreas or liver transplant and exposed to gadolinium contrast agents.
  Interventions: Drug: Gadolinium contrast dye
- Non-transplant patients, MRI with Gadolinium contrast dye: Non-transplant patients exposed to gadolinium contrast.
  Interventions: Drug: Gadolinium contrast dye
- Healthy controls, no transplant no Gadolinium contrast dye: Age- and sex-matched healthy controls not exposed to gadolinium contrast.

INTERVENTIONS:
Drug: Gadolinium contrast dye — Gadolinium contrast dye administered during MRI
  Groups: Non-transplant patients, MRI with Gadolinium contrast dye; Transplant patients, MRI with Gadolinium contrast dye

SUMMARY:
Gadolinium contrast agents are frequently administered for MRI imaging. Very little is known of its toxicity outside of patients with reduced renal function.

DETAILED DESCRIPTION:
Gadolinium contrast is administered to patients during MRI imaging. Recently, the investigators have observed potential gadolinium toxicity in some patients. To investigate this, the investigators propose to collect clinical data and lab data obtained as a part of clinical care. The investigators also plan to obtain 25 cc of peripheral blood at 2-4 weeks, 4-6 weeks and again at 3 months to identify unique monocyte signatures, gene polymorphisms, and to quantitate circulating fibrocytes (in fresh blood and after culture). Plan to enroll 15 patients with kidney, pancreas or liver transplant and exposed to gadolinium contrast agents, 15 non-transplant patients exposed to gadolinium contrast and 30 age- and sex-matched healthy controls not exposed to gadolinium contrast.

ELIGIBILITY:
Inclusion Criteria:

* Renal, pancreas or liver transplant OR those without organ transplant OR controls
* Age 18-70
* Both gender
* Exposure to gadolinium contrast agents (no exposure in controls)
* Have had a transplant, have had a contrast dye with an MRI
* Have not had a transplant and have had a contrast dye with an MRI
* Healthy person who has not had an MRI or gadolinium for any other reason.

Exclusion Criteria:

* End stage kidney disease or Stage 5
* Previous diagnosis of Nephrogenic Systemic Fibrosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Gadolinium exposed patients. We will use age- and sex-matched controls with and without organ transplants and not exposed to gadolinium contrast agents (within the last 3 years) as controls.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
total number of circulating fibrocytes | 2-4 weeks
  2-4 weeks after gadolinium contrast exposure

CONTACTS AND LOCATIONS:
Overall Officials: Sundararaman Swaminathan, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States